CLINICAL TRIAL: NCT01450449
Title: A Randomized Phase III Study of Short Course (One-week) Radiation Therapy Versus Standard Course (Three-week) Radiation Therapy in Elderly and/or Frail Patients With Newly Diagnosed Glioblastoma Multiforme
Brief Title: Short Course vs. Standard Course Radiotherapy in Elderly and/or Frail Patients With Glioblastoma Multiforme
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: International Atomic Energy Agency (Other Government)
Collaborators: Fundación Escuela de Medicina Nuclear (Other); N.N. Alexandrov National Cancer Centre (Other Government); Hospital A.C. Camargo (Other); Irmandade Santa Casa de Misericórdia de Porto Alegre (Other); Instituto de Radiomedicina (IRAM) (Unknown); Post Graduate Institute of Medical Education and Research, Chandigarh (Other); Dr Cipto Mangunkusumo General Hospital (Other); Maria Sklodowska-Curie National Research Institute of Oncology (Other); Chiang Mai University (Other); Salah Azaïz Cancer Institute (Other); Wilson Roa Professional Corporation (Unknown); Cancer Trials Ireland (Network); Ege University (Other); High Technology Medical Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E33033
Record Dates: First submitted 2011-10-10; First posted 2011-10-12 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Glioblastoma Multiforme
Keywords: GBM, fractionation, short course, standard course
MeSH Terms: conditions — Glioblastoma | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 - Short Course Radiotherapy (Experimental): Short Course
  Interventions: Radiation: Radiotherapy
- Arm 2 - Standard Course Radiotherapy (Active Comparator): Standard Course
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Radiation: Radiotherapy — 25 Gy in 5 daily fractions over 1 week
  Arms: Arm 1 - Short Course Radiotherapy
Radiation: Radiotherapy — 40 Gy in 15 daily fractions over 3 weeks
  Arms: Arm 2 - Standard Course Radiotherapy

SUMMARY:
This is a multi-centre prospective, non-inferiority trial. Patients will be randomized to two treatment groups in a 1:1 ratio and will be stratified by age, Karnofsky Performance Status and extent of the surgical resection.

This study will assess the effect of a one-week radiotherapy regimen in comparison with a three-week radiotherapy regimen on the survival of elderly and/or frail patients with glioblastoma multiforme (Frail: ≥>50 years old and with a KPS of 50% or less50%-70%; Elderly and frail: ≥65 years and with a KPS of 50% - 70%; Elderly: ≥65 years and with a KPS of 80% - 100%).

DETAILED DESCRIPTION:
This is a multi-centre prospective, non-inferiority trial. Patients will be randomized to two treatment groups in a 1:1 ratio and will be stratified by:

* Age (<65 and ≥65 years old)
* Karnofsky Performance Status (≤70 and > 7050 or higher)
* Extent of the resection at surgery (biopsy only versus complete/near total and gross total or incomplete /partial resection)

Randomization:

Patients will be randomized to receive one of the two following treatments:

Arm 1:

* Short Radiotherapy
* 25 Gy/5 fractions
* 1 week (5 fractions per week)

Arm 2:

* Regular Radiotherapy
* 40 Gy/15 fractions
* 3 weeks (5 fractions per week)

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed newly diagnosed glioblastoma multiforme (GBM, WHO grade IV). The histological diagnosis must have been made locally after biopsy or neurosurgical tumour resection.
* Initial surgery/biopsy at diagnosis performed < 6 weeks (42 days) prior to randomization.
* Patient's age is 50 years or older.
* Karnofsky performance status is 50% or higher.
* Patients may have received and continue to receive corticosteroids, but they have to be on a stable or decreasing dose for at least 14 days prior to randomization.
* Patients must not have received prior chemotherapy or radiotherapy.
* Patient is able (i.e. sufficiently fluent) and willing to complete the quality of life questionnaires in either English or any other language the questionnaire is officially translated into. The baseline assessment (prior to start of radiotherapy) must already have been completed. Inability (illiteracy, loss of sight, or other equivalent reason) to complete the questionnaires will not make the patient ineligible for the study. In centres where patients are not able to read or write, proxy interviews will be conducted in-person or via telephone by the nurse at that particular centre.
* Patient consent must be obtained according to local institutional policy. It will be the responsibility of the local participating investigators to obtain the necessary local clearance, and to indicate in writing to the IAEA Study Coordinator that such clearance has been obtained, before the trial can commence in that centre. A copy of the initial full board ERB approval and approved consent form must be sent to the Project Officer at IAEA. The patient must sign the consent form prior to randomization or registration.
* Patients must be accessible for treatment and follow-up. Investigators must assure themselves the patients randomized on this trial will be available for complete documentation of the treatment, adverse events, and follow-up.
* Protocol treatment is to begin within 2 weeks of patient randomization.

Exclusion Criteria:

* Patients with a history of other malignancies, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumours curatively treated with no evidence of disease for 3 or more years.
* Patients with a serious active infection or other serious underlying medical conditions that would impair the ability of the patient to receive protocol treatment or comply with protocol.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2009-02; Primary Completion 2013-12 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 2.5 years
  The time from randomization to the time of death from any cause.

SECONDARY OUTCOMES:
Progression-free survival | 2.5 years
  2.5 years including six months of follow-up after initial accrual.
Quality of Life | 2.5 years
  Quality of life will be assessed prior to study randomization and 4 weeks following completion of radiotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Elena Fidarova, Principal Investigator — International Atomic Energy Agency
Locations (15):
- Fundacion Escuela de Medicina Nuclear, Mendoza, Argentina
- N.N. Alexandrov National Cancer Centre of Belarus, Minsk, Belarus
- Brazil (2):
  - Irmandade de Santa Casa de Misericordia de Porto Alegre, Porto Alegre
  - Hospital "A.C. Camargo", Fundacao "Antonio Prudente", São Paulo
- Wilson Roa Professional Corporation, Edmonton, Canada
- Instituto de Radiomedicina (IRAM), Santiago, Chile
- Regionaalhailga, Tallinn, Estonia
- High Technology Medical Center, University Clinic, Tbilisi, Georgia
- Postgraduate Institute of Medical Education and Research (PGIMER), Chandigarh, India
- Cipto Magunkusumo General Hospital, University of Indonesia, Jakarta, Indonesia
- ICORG The All Ireland Cooperative Oncology, Dublin, Ireland
- Marie Curie- Sklodowska Institute of Oncology, Warsaw, Poland
- Division of Therapeutic Radiology and Oncology, Faculty of Medicine, Chiang Mai University, Chiang Mai, Thailand
- Institut National de Cancer Salah Aziz, Ministere de la Sante Publique, Tunis, Tunisia
- Ege University Hospital, Izmir, Turkey (Türkiye)

REFERENCES:
- [Background] Newall J, Ransohoff J, Kaplan B. Glioblastoma in the older patient: how long a course of radiotherapy is necessary? J Neurooncol. 1988 Dec;6(4):325-7. doi: 10.1007/BF00177427. PMID 2851647
- [Background] Bauman GS, Gaspar LE, Fisher BJ, Halperin EC, Macdonald DR, Cairncross JG. A prospective study of short-course radiotherapy in poor prognosis glioblastoma multiforme. Int J Radiat Oncol Biol Phys. 1994 Jul 1;29(4):835-9. doi: 10.1016/0360-3016(94)90573-8. PMID 8040031
- [Background] Kleinberg L, Slick T, Enger C, Grossman S, Brem H, Wharam MD Jr. Short course radiotherapy is an appropriate option for most malignant glioma patients. Int J Radiat Oncol Biol Phys. 1997 Apr 1;38(1):31-6. doi: 10.1016/s0360-3016(97)00222-8. PMID 9212001
- [Background] Jeremic B, Shibamoto Y, Grujicic D, Milicic B, Stojanovic M, Nikolic N, Dagovic A, Aleksandrovic J. Short-course radiotherapy in elderly and frail patients with glioblastoma multiforme. A phase II study. J Neurooncol. 1999 Aug;44(1):85-90. doi: 10.1023/a:1006356021734. PMID 10582674
- [Background] Roa W, Brasher PM, Bauman G, Anthes M, Bruera E, Chan A, Fisher B, Fulton D, Gulavita S, Hao C, Husain S, Murtha A, Petruk K, Stewart D, Tai P, Urtasun R, Cairncross JG, Forsyth P. Abbreviated course of radiation therapy in older patients with glioblastoma multiforme: a prospective randomized clinical trial. J Clin Oncol. 2004 May 1;22(9):1583-8. doi: 10.1200/JCO.2004.06.082. Epub 2004 Mar 29. PMID 15051755
- [Derived] Roa W, Kepka L, Kumar N, Sinaika V, Matiello J, Lomidze D, Hentati D, Guedes de Castro D, Dyttus-Cebulok K, Drodge S, Ghosh S, Jeremic B, Rosenblatt E, Fidarova E. International Atomic Energy Agency Randomized Phase III Study of Radiation Therapy in Elderly and/or Frail Patients With Newly Diagnosed Glioblastoma Multiforme. J Clin Oncol. 2015 Dec 10;33(35):4145-50. doi: 10.1200/JCO.2015.62.6606. Epub 2015 Sep 21. PMID 26392096